CLINICAL TRIAL: NCT06853444
Title: A Phase 1/2 Study on the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Efficacy of the Anti-BAFF-R Monoclonal Antibody, ESG206, in Patients With Primary Immune Thrombocytopenia (ITP)
Brief Title: A Phase 1/2 Study of ESG206 in Patients With Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Escugen Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESG206-ITP-01
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-02

CONDITIONS: Immune Thrombocytopenia (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ESG206 dose level 1 (Experimental): ESG206 will be administered intravenously at dose level 1.
  Interventions: Drug: ESG206
- ESG206 dose level 2 (Experimental): ESG206 will be administered intravenously at dose level 2.
  Interventions: Drug: ESG206
- ESG206 dose level 3 (Experimental): ESG206 will be administered intravenously at dose level 3.
  Interventions: Drug: ESG206
- ESG206 dose level 4 (Experimental): ESG206 will be administered intravenously at dose level 4.
  Interventions: Drug: ESG206

INTERVENTIONS:
Drug: ESG206 — Administered via intravenous (IV) infusion
  Other Names: ESG206-2
  Arms: ESG206 dose level 1
Drug: ESG206 — Administered via intravenous (IV) infusion
  Arms: ESG206 dose level 2
Drug: ESG206 — Administered via intravenous (IV) infusion
  Arms: ESG206 dose level 3
Drug: ESG206 — Administered via intravenous (IV) infusion
  Arms: ESG206 dose level 4

SUMMARY:
This is a multicenter, open-label Phase1/2 study aimed at evaluating the safety, tolerability, pharmacokinetic (PK) profile, pharmacodynamics (PD), immunogenicity, and preliminary efficacy of ESG206. The study will be conducted in patients with primary immune thrombocytopenia.

DETAILED DESCRIPTION:
Phase 1 is a dose escalation study, and Phase 2 is an extended cohort study, subjects will be treated with ESG206.

In Phase 1&2, the study includes Screening (no more than 28 days), Treatment (14 weeks), and the post-treatment follow-up (8 weeks), for those sufferring a treatment failure, the safe follow-up will be conducted 28 days after the last dose.

And the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary efficacy of ESG206 in primary ITP will be assessed in this study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Willing and able to provide written informed consent for this trial.
* 2. Male or female, age ≥ 18 years on the day of signing the informed consent form.
* 3. Diagnosed with primary immune thrombocytopenia (ITP), and having received treatment of corticosteroids ± intravenous immunoglobulin (IVIG) in the past.
* 4. At the time of the last ITP treatment, loss of response, insufficient response, no response or intolerance occurred.
* 5. At screening, Platelet Count revealed < 30 * 10^9/L twice (with an interval of at least 24 hours between the two tests).
* 6. Subjects must have adequate organ function.
* 7. The World Health Organization (WHO) bleeding scale is 0-1.
* 8. Fertile men and women of reproductive age must agree to use effective contraception from the time they sign the informed consent until 180 days after the last dose of the trial drug. Women of reproductive age include premenopausal women and women within 2 years after menopause. Women who are fertile must have a pregnancy test within 7 days before the trial drug is first given and the result should be negative.

Exclusion Criteria:

* 1. Diagnosed with secondary immune thrombocytopenia, or there is evidence that the patient has a secondary cause of immune thrombocytopenia, or the patient has multiple immune cytopenias.
* 2. Previously received B-cell depletion therapy (e.g., rituximab, Ianalumab, etc.).
* 3. Received platelet transfusion or whole blood transfusion, plasma exchange, or any other rescue treatment within 14 days before the first administration of the trial drug.
* 4. Participated in other investigational drug clinical studies within 4 weeks before the first administration of the investigational drug or within 5 half-lives of the investigational drug received (whichever is longer).
* 5. Underwent splenectomy within 12 weeks before the first administration of the investigational drug.
* 6. Received traditional Chinese medicine treatment with definite platelet-raising effects within 1 week before the first administration of the trial drug.
* 7. Underwent major surgery within 4 weeks before the first administration of the investigational drug or needs to undergo major elective surgery during the study period.
* 8. Diagnosed with Evans syndrome or any other cytopenia (patients with mild anemia related to bleeding or iron deficiency are eligible for inclusion in the study).
* 9. Patients with current or previous life-threatening bleeding related to thrombocytopenia.
* 10. Patients with concurrent coagulation disorders and/or receiving antiplatelet or anticoagulant therapy (e.g., warfarin, clopidogrel, or new oral anticoagulants), except for low-dose acetylsalicylate (≤150 mg/day).
* 11. Patients with deep vein thrombosis or arterial thrombosis within 6 months before enrollment, and/or with risk factors for hereditary thrombophilia.
* 12. Patients with a history of severe cardiovascular and pulmonary diseases.
* 13. Patients with uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg).
* 14. Patients with human immunodeficiency virus (HIV) infection, or active hepatitis B or C, or liver cirrhosis.
* 15. Patients with active viral, bacterial, or other infections requiring systemic treatment during the screening period, or with a history of clinically significant recurrent infections (e.g., bacterial infection with capsule). Patients with a history of tuberculosis (TB) or latent TB who have undergone anti-TB treatment may be eligible for inclusion.
* 16. Patients who received live or attenuated live vaccines within 4 weeks before the first administration of the investigational drug.
* 17. Patients with a history of or current malignant tumors, except for cured non-melanoma skin cancer, carcinoma in situ (e.g., cervical cancer, breast cancer, bladder cancer, prostate cancer), and cancers that have been in complete remission for at least 3 years without evidence of recurrence.
* 18. Patients with any severe and/or unstable pre-existing medical, mental, or other conditions that the investigator deems may interfere with the patient's efficacy, safety, informed consent, or compliance with the study procedures.
* 19. Patients with known immediate or delayed hypersensitivity reactions to monoclonal antibodies or components of the trial drug, or with a history of allergic constitution.
* 20. Pregnant or lactating women.
* 21. Patients who are unwilling or unable to follow the protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Any Treatment Emergent Adverse Events and Serious Treatment Emergent Adverse Events | Up to 24 weeks.
  Treatment-emergent adverse events (TEAEs) were defined as: Any adverse event (AE) that happens after treatment initiation, or AE that was present at time of treatment initiation but worsened after treatment initiation, or AE that was present and resolved prior to treatment and reappeared after treatment initiation after the start of study drug through 28 days after the last dose of study drug or the last post-treatment follow-up. The severity was graded based on the National Cancer Institute's Common Terminology Criteria for Adverse Events.
Confirmed response rate | Between Week 1 Day 1 and Week 25 Day 1
  Confirmed response is defined as a platelet count of equal or above 50 G/L at two (or more) consecutive assessments at least 7 days apart, in the absence of:
  Rescue treatment for ≥4 weeks prior to the assessment of the platelet count, and New immune thrombocytopenia (ITP) treatment before reaching a confirmed response.

SECONDARY OUTCOMES:
AUC0-inf | up to Week 25
  Area under the serum concentration time curve (AUC) from time 0 extrapolated to infinity
Cmax | up to Week 25
  Maximum observed plasma concentration
Tmax | up to Week 25
  Time to maximum plasma concentration
T1/2 | up to Week 25
  Half-life
Response rate at each timepoint | Between Week 1 Day 1 and Week 25 Day 1
  Percentage of participants with a platelet count of at least 50 G/L in the absence of rescue treatment/new ITP treatment.
Complete Response rate at each timepoint | Between Week 1 Day 1 and Week 25 Day 1
  Percentage of participants with a platelet count of at least 100 G/L in the absence of rescue treatment/new ITP treatment.
Best Response rate at each timepoint | Between Week 1 Day 1 and Week 25 Day 1
  Percentage of participants with Response or Complete Response in the absence of rescue treatment/new ITP treatment.
Time to confirmed response | Between Week 1 Day 1 and Week 25 Day 1
  Time from the first administration of ESG206 to the first assessment in the first sequence of two (or more) platelet assessments meeting the criteria of a confirmed response as defined by the primary endpoint.
Time to complete response | Between Week 1 Day 1 and Week 25 Day 1
  Time from the first administration of ESG206 to the first assessment meeting the criteria of a complete response.
Time to treatment failure | Between Week 1 Day 1 and Week 25 Day 1
  Time from the first administration until platelet count below 30 G/L, need for a rescue treatment or start of a new therapy or death.
Duration of response | Between Week 1 Day 1 and Week 25 Day 1
  Time from achievement of response to loss of response
Duration of complete response | Between Week 1 Day 1 and Week 25 Day 1
  Time from achievement of complete response to loss of complete response.
Percentage of participants receiving rescue treatment | Between Week 1 Day 1 and Week 25 Day 1
  Assess the need of rescue treatment by percentage.
Change from baseline in absolute number of CD19+ B cell counts | Between Week 1 Day 1 and Week 25 Day 1
  Post baseline absolute number of CD19+ B cell counts compare with baseline
Change from baseline in absolute number of CD20+ B cell counts | Between Week 1 Day 1 and Week 25 Day 1
  Post baseline absolute number of CD20+ B cell counts compare with baseline
Incidence of anti-drug antibodies in serum (ADA assay) over time | Between Week 1 Day 1 and Week 25 Day 1
  Anti-drug antibodies (ADA) will be evaluated in samples collected from all participants assess the immunogenicity of ESG206

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No